CLINICAL TRIAL: NCT01975597
Title: Pilot Study of Bone Biopsy and Aspirate in Women With Metastatic Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: held for blocking amendment then determined not to re-open
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2013.053; HUM00075575 (Other: University of Michigan)
Record Dates: First submitted 2013-09-03; First posted 2013-11-04 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow, peripheral blood, tumor tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bone marrow aspirates and biopsy
  Interventions: Procedure: Bone marrow aspirates and biopsy

INTERVENTIONS:
Procedure: Bone marrow aspirates and biopsy

SUMMARY:
This is a feasibility study to demonstrate the team's ability to collect bone marrow aspirates and biopsies for research purposes from women with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic breast cancer (any site) age 21 or older
* Patients willing and able to provide informed consent & perform study procedures
* Patients may enroll with recently (with 2 months) progressive tumor burden
* Performance status of 0,1 or 2

Exclusion Criteria:

* Patients unable or unwilling to provide informed consent and or perform study procedures
* Patients with active, uncontrolled coagulopathy
* Patients on treatment dose anticoagulation or an International Normalised Ratio of 2 or greater if on warfarin
* Patients who are known to be pregnant are not eligible to participate in this study during the time of the pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are receiving care for metastatic breast cancer at University of Michigan Rogel Cancer Center will be recruited for this study to donate samples.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11-19 (Actual); Study Completion 2014-11-19 (Actual)

PRIMARY OUTCOMES:
Number of patient that agree to undergo 2 biopsy's strictly for research purposes. | At 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Van Poznak, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States